CLINICAL TRIAL: NCT01252316
Title: An In-Hospital VSI CPR Dissemination Study Using Nurses and Volunteers
Brief Title: Cardiopulmonary Resuscitation (CPR) Dissemination Study Using Nurses and Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CRS-812096
Record Dates: First submitted 2010-11-29; First posted 2010-12-02 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2015-12

CONDITIONS: Cardiovascular Risk Factors; Coronary Disease; Cardiac Arrest
MeSH Terms: conditions — Coronary Disease; Heart Arrest

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard CPR (Active Comparator): Individuals will learn the Standard form of CPR (30:2, compressions:breathes) Main data points being collected at various increments over 12 months are: 1) Comfort Level with using CPR 2) Secondary Training "multiplier effect" 3) CPR Skills
  Interventions: Other: CPR Training using the Family and Friends CPR Anytime VSI Kit
- Recruitment with Volunteers (Active Comparator): UPHS volunteer subjects will be identified by hospital stakeholders, and they will be given surveys to assess their confidence, attitudes and beliefs towards this program at 3-month integrals.
  Interventions: Other: Implementation of an In-Hospital CPR Training Model
- Recruitment with Nurses (Active Comparator): UPHS Nurse subjects will be identified by hospital stakeholders, and they will be given surveys to assess their confidence, attitudes and beliefs towards this program at 3-month integrals.
  Interventions: Other: Implementation of an In-Hospital CPR Training Model
- Chest Compressions Only CPR (Active Comparator): Individuals will learn the chest compression only form of CPR (no rescue breathes) Main data points being collected at various increments over 12 months are: 1) Comfort Level with using CPR 2) Secondary Training "multiplier effect" 3) CPR Skills
  Interventions: Other: CPR Training using the Family and Friends CPR Anytime VSI Kit

INTERVENTIONS:
Other: CPR Training using the Family and Friends CPR Anytime VSI Kit — Subjects will be trained using the American Heart Association's Family and Friends CPR Anytime Kit. The subject's will undergo training in-hospital then they will be encouraged to take the kit home with them to practice CPR with their family members and friends.
  Arms: Chest Compressions Only CPR; Standard CPR
Other: Implementation of an In-Hospital CPR Training Model — UPHS Nurses and Volunteers will be trained in our in-hospital CPR Training Model using VSI Kits, and encouraged to implement the training program in their respective hospitals.
  Arms: Recruitment with Nurses; Recruitment with Volunteers

SUMMARY:
Each year in the United States, 300,000 people suffer from Cardiac Arrest (CA), and of them there is a 90% mortality rate. Out-of-Hospital arrests in particular have a 1-5% survival to hospital discharge. High quality CPR is crucial to lowering the mortality rate and increasing survival, yet only 15-30% of out-of-hospital CA victims receive bystander CPR. Studies have shown that prompt administration of CPR dramatically improves outcomes. In a recent study from Switzerland, lay bystander CPR doubled the survival rate at one month. Our study will look to train family members of at-risk cardiac patients in the skills of CPR through the American Heart Associations (AHA) CPR Anytime Friends and Family Personal Learning Program (CPR Anytime) to see if these family members are able to learn and perform quality CPR in the event that their family member should suffer a cardiac arrest. The unique feature of the CPR Anytime training is that it is a low-cost, self-learning, video-based program that can be completed in under 30 minutes, saving the time and expense of traditional CPR training courses. While initial work has proven that teaching CPR in hospital using the VSI kit is feasible, little research has been conducted to make the program sustainable.

DETAILED DESCRIPTION:
The long term goal of our work is to implement real world CPR training strategies that match training locales with at-risk populations, maximize resuscitation skill retention, and promote willingness to act. To accomplish this, we will empower stakeholders at UPHS hospitals to develop local implementation approaches, using either UPHS volunteers or nursing staff as VSI proctors. These stakeholders will be studied as a research subset. The VSI proctors will use the AHAs CPR Anytime kit, and will work with family members of patients at high risk for a CA to learn lifesaving CPR skills. We will use a modified AHA CPR video using the new AHA recommendations for bystanders which suggests doing chest compression only CPR. Using the original AHA video and the modified chest compression only video, we will randomize family members of patients at high risk for CA to one of these groups. The VSI proctors will also be blinded to which video these subjects will be watching. We will follow up with the family members at 1 month, 3 months, 6 months and 12 months to see if they retained their CPR knowledge and skills and to see if they had been in a situation where their CPR skills were needed and assess whether they performed their skills or not. We will also measure the number of people with whom the subjects shared their CPR Anytime kits a quantity known as the multiplier effect to determine if they had shared the CPR Anytime kit with their family and friends, thereby increasing the possible number of lay persons trained in CPR and in turn able to perform bystander CPR if needed. We will also assess the perceptions and attitudes of the nurses and volunteers regarding this project.

ELIGIBILITY:
Inclusion Criteria:

* Family Member's of Patients with known coronary disease or cardiovascular risk factors, such as history of diabetes and hypertension.

Exclusion Criteria:

* If someone is physically unable to undergo CPR Training
* Someone who has received CPR training in the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Assessing Nurses and Volunteers implementation of the in-hospital CPR Training Program | 2 years
  To determine if volunteers or nursing staff can adequately implement a CPR Training Program for at risk family members of patients hospitalized for cardiac risk-factors. Subjects will be given "enroller surveys" in 3-month integrals to assess comfort level with the program.

SECONDARY OUTCOMES:
CPR Skills Performance and Retention | up to 1 year
  To assess skill performance by subject family members and retention with chest compression only CPR versus standard CPR education. Subjects will be asked to perform 2 minutes of CPR on a Laerdal SkillReporter ResusciAnne mannequin.
Assessing bystander CPR training dissemination | up to 1 year
  To quantify the multiplier effect, an assessment of the number of people who received secondary CPR training via CPR Anytime kits shared with them by study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S Abella, MD, MPhil, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania